CLINICAL TRIAL: NCT07188493
Title: Analysis and Evaluation of the Effectiveness of Remote Rehabilitation Using a Knee Brace in People With Degenerative Disease
Brief Title: Remote Rehabilitation With Knee Brace for Individuals With Degenerative Joint Disease
Acronym: JC3D
Status: Active, not recruiting | Type: Observational
Sponsor: MDH sp. z o.o. (Industry)
Collaborators: Sporto Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: JC3D/2024
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis (OA); Joint Diseases; Knee Brace
Keywords: OA; orthosis; telerehabilitation; knee brace; knee; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Participants in this group follow a complete telerehabilitation protocol, including:
  * An individually tailored home-based kinesitherapy program delivered through the Qmed Play mobile application
  * A custom-made rehabilitation knee brace (Jointcraft 3D Knee Brace with range-of-motion adjustment, MDH sp. z o.o., Maratońska 104, 94-007 Łódź, Poland) integrated with motion sensors (Qmed Sensors, MDH sp. z o.o., Maratońska 104, 94-007 Łódź, Poland) and the Qmed Play mobile application
- Group B: Participants in this group receive:
  * An individually tailored home-based kinesitherapy program
  * A custom-made rehabilitation knee brace (Jointcraft 3D Knee Brace with range-of-motion adjustment, MDH sp. z o.o., Maratońska 104, 94-007 Łódź, Poland)
- Group C: Participants in this group receive:
  * An individually tailored home-based kinesitherapy program
  * A standard functional knee brace (Follow Force Knee Brace with range-of-motion adjustment, MDH sp. z o.o., Maratońska 104, 94-007 Łódź, Poland)

SUMMARY:
The goal of this observational study is to learn how well remote rehabilitation and offloading the inner part of the knee joint using a custom-made knee brace work as non-surgical treatments for people with unicompartmental knee osteoarthritis.

The main question it aims to answer is:

Does the remote rehabilitation system improve symptoms and function in people with knee osteoarthritis?

Researchers will compare three groups of participants to see how different types of knee braces and rehabilitation methods affect outcomes:

Group A will use a custom-made knee brace connected to a mobile app and motion sensors.

Group B will use a custom-made knee brace daily and perform prescribed exercises.

Group C will use a standard off-the-shelf functional knee brace daily and perform the same prescribed exercises.

Participants will:

Wear their assigned brace for 6 months

Complete surveys (VAS, KOOS, and Laitinen)

Have their knee range of motion and body weight measured

ELIGIBILITY:
Inclusion Criteria:

* Unicompartmental knee osteoarthritis (medial compartment), Kellgren-Lawrence grade I-III, confirmed by imaging; affecting one lower limb (with predominant symptoms in either the right or left leg)
* Age between 45 and 75 years
* Preserved passive knee extension; flexion contracture of up to 20 degrees of extension deficit is acceptable
* Signed informed consent for participation in the clinical investigation

Exclusion Criteria:

* Bicompartmental knee osteoarthritis with similar symptom severity in both compartments
* Neurological disorders
* Rheumatoid arthritis
* Coexisting dysfunctions of the hip and/or ankle joint of the affected limb
* Ligament injuries (ACL, PCL, MCL, LCL) and/or meniscus injuries (medial or lateral) causing significant joint instability (moderate instability due to ligament insufficiency, common in osteoarthritis, is not excluded)
* Bone fractures
* Sensory disturbances in the lower limbs
* Passive knee extension deficit greater than 20 degrees
* Major surgical procedures involving the knee joint within the last 6 months
* Lack of informed consent and/or inability to establish reliable verbal-logical communication with the participant
* Other medical conditions preventing independent application of the brace and/or use of the mobile application

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be observed from patients receiving conservative treatment for medial compartment knee osteoarthritis at the Sporto Clinic. The study population includes adults aged 45 to 75 years diagnosed with unicompartmental knee osteoarthritis (Kellgren-Lawrence grade I-III) in one lower limb, confirmed by imaging. Participants are community-dwelling individuals able to follow a home-based exercise program and use a functional knee brace.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
KOOS Questionnaire (Knee injury and Osteoarthritis Outcome Score) | At first and final visit (6 months)
  The KOOS questionnaire is a validated and internationally recognized self-reported tool, officially translated into Polish, used to assess knee-related symptoms. It consists of five subscales: pain, knee stiffness, daily living function, sports and recreational activity, and knee-related quality of life.
  The maximum score of 100 indicates no symptoms or limitations, while a score of 0 indicates extreme symptom severity.
VAS Scale (Visual Analog Scale) | At first and final visit (6 months)
  A subjective scale for evaluating pain intensity. This 10-point scale measures how strong the participant's pain is, where 1 means no pain and 10 means unbearable pain.
Laitinen Scale | At first and final visit (6 months)
  A subjective, point-based tool assessing pain based on four features: intensity, frequency, use of pain medication, and physical activity limitation.
  Each category is scored from 0 to 4, where 0 means no issue, and 4 indicates the most severe problem.
Lower Limb Ortogram | At first and final visit (6 months)
  Anteroposterior (AP) radiograph of both lower limbs taken in a standing position, with feet hip-width apart and in a neutral position.
  Measurements include the angle between the mechanical axis of the femur and tibia, and the medial joint space width (JSW) of the knee [mm].
Range of Motion (ROM) of the Knee Joint | At first and final visit (6 months)
  Angular measurement of the knee's flexion and extension using an electronic goniometer.
  For flexion: the patient lies on their back with legs extended; the goniometer axis is placed at the lateral femoral epicondyle, with the fixed arm aligned with the greater trochanter and the movable arm following the lateral malleolus as the patient actively bends the knee.
  For extension: the patient lies face down with legs bent at the knees, positioned so that the knees extend beyond the edge of the examination table to allow full extension or hyperextension. Goniometer placement follows the same protocol.
  Measurements are taken for both limbs.
Custom Satisfaction Questionnaire | At the final visit (6 months)
  A proprietary survey assessing patient satisfaction with the telerehabilitation program, as well as comfort and perceived effectiveness of the cage-type knee brace used in the conservative treatment of knee osteoarthritis. The survey is based on a 5-point scale, where 1 represents a poor outcome, 5 indicates an excellent result, and 3 denotes no change.

SECONDARY OUTCOMES:
BMI (Body Mass Index) | At first and final visit (6 months)
  BMI is calculated as weight [kg] divided by height squared [m²]. It is considered a significant risk factor in the severity and progression of knee osteoarthritis.
  A simplified BMI classification is used in this study:
  <18.5 - underweight; 18.5-24.99 - normal; >24.99 - overweight
Lower Limb Circumference Measurements | At first and final visit (6 months)
  Circumference measurements (in cm) of the thigh (10 cm above mid-patella), knee (at mid-patella), and calf (15 cm below mid-patella) on both braced and non-braced limb; used for asymmetry assessment, monitoring changes over time, and brace sizing.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Domżalski, M.D., Principal Investigator — Sporto
Locations (1):
- Sporto, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves a small, single-center population, and the data include potentially identifiable medical and imaging information. The data are intended for internal analysis and publication in aggregate form only.